CLINICAL TRIAL: NCT05842135
Title: REsectability Small Bowel Obstruction LAParoscopic (RESBOLAP) Score. Multicentric Data Registry
Acronym: RESBOLAP
Status: Completed | Type: Observational
Sponsor: San Salvatore Hospital, AST Pesaro-Urbino (Other)
Responsible Party: Principal Investigator, Diego Coletta, Principal Investigator, San Salvatore Hospital, AST Pesaro-Urbino
Other Study IDs: CERP22078
Record Dates: First submitted 2023-04-11; First posted 2023-05-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-04

CONDITIONS: Small Bowel Obstruction
Keywords: indocyanine green fluorescence; small bowel obstruction; fluorescent angiography; resectability score; laparoscopic emergency surgery

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic approach to small bowel obstrcuction — Bowel viability assessment by indocyanine green fluorescent angiography during laparoscopic approach to small bowel obstruction
  Other Names: indocyanine green fluorescent angiograhy

SUMMARY:
AIM OF THE STUDY The aim of the study is to develop a Resectability Laparoscopic Score as a helpful instrument during intraoperative decision-making in the setting of emergency laparoscopic surgery for small bowel obstruction (SBO) by analyzing a multicenter data registry.

DESIGN OF THE STUDY This is a multicenter study composed of a first phase of prospective data collection from patients that undergo laparoscopic surgery with a diagnosis of SBO and undergo Indocyanine green (ICG) fluorescence angiography (FA) for doubts about bowel viability after the resolution of the obstructive mechanism; the second phase of retrospective analysis to develop the Resectability Score.

METHODS The FA should be performed in all patients undergoing laparoscopic surgery for SBO that presents concerns bowel viability after the resolution of the occlusive mechanism, with consequent intraoperative enrolment in the study Registry.

The investigators adopted the modified Bulkley classification of the fluorescent patterns to identify which patients need more FA to assess bowel vitality.

It is expected that most patients for whom the FA will be performed are those with patterns 2 or 3, representing the study's primary object.

All participant centers must adopt the same technique to perform FA with the attempt to homogenize the procedure.

Twenty-five milligrams of ICG powder is suspended in 10 ml of sterile water and administered intravenously through a peripheral vein and in small repeatable boluses of 2 ml in order to evaluate the intestinal microcirculation extemporaneously. The presence and pattern of arterial supply is tested and compared with that of healthy bowel. Proper clearance of the dye was also appraised to verify adequate venous drainage. Following the reversal of the underlying cause of the ischaemic injury, and after generous irrigation with warm saline, the involved bowel segment was further evaluated with FA after 10 min, regardless of the return of visible peristalsis.

Routine postoperative clinical judgment will be considered sufficient to check bowel vitality.

The need for a second-look surgery and delayed resections will be recorded. All centers could participate with a maximum of 3-4 members (co-authorship) Data will be recorded by a simple and brief online Case Report Form (CRF) on which upload also a photo/brief video of the FA, will be filled out by every participating center for each patient.

A link to a Google Form and the necessary documents will be sent to every center after they have accepted to participate in the study.

DETAILED DESCRIPTION:
Albeit the role of laparoscopy in the treatment of acute small bowel obstruction (SBO) has grown significantly over the last decade, the inability to obtain an adequate evaluation of compromised bowel segments has been considered as real limitation. This is essentially due to a reduced field of view owing to intestinal distension, the minimized haptic feedback obtained and limited bi-dimensional visualization. As a consequence, the presence of normal visual clues to irreversible vascular insufficiency is much reduced.

Such signs include stable discoloration of the bowel wall, absence of peristaltic movements and apparent mesenteric pulsation. Intestinal perfusion and viability are largely assessed by means of the clinical eye. However, this method lacks objectivity and accuracy, irrespective of a surgeon's experience. Routinely clinical judgment may be appropriate, but the rate of conversion due to concerns regarding bowel viability can be high. Where there are concerns for intestinal ischaemic injury without absolute indications to bowel resection (areas of mural gangrene or bowel necrosis with perforation) intestinal compromise can be appraised by real-time fluorescent analysis of the vascular supply.

Some authors reported their experience on the use of the ICG fluorescent angiography (FA) to assess bowel viability during laparoscopic approach in emergency surgery for SBO, with promising results. Nowadays, an important drawback of qualitative intraoperative assessment of bowel compromise with FA is the interpretation and definition of the boundaries between bowel viability and irreversible ischemia in order to avoid or reduce the rate of delayed bowel necrosis and perforation. An instrument more objective as possible to help surgeons during the intraoperative decision-making is lacking. A resectability score could be resolutive but a large amount of data from a multicentric data registry is needed.

Finally, when the registry will be completed, a logistic regression analysis will be used to identify independent predictive factors of bowel resectability by calculation of odds ratios and its 95% CI based on delayed bowel resection rate too. Significant continuous variables will be transformed into categorical variables using receiver operating characteristic (ROC) curves. The sample size required for the development of the Score was determined according to previous reports. The number of unnecessary bowel resections has been estimated around 46%. Two studies on ICG-fluorescence angiography use during laparoscopic surgery for SBO reported 28.6% of resection rate. The investigators adopted this degree of difference as the maximum error tolerance of 17.4%. Considering a power of 0.9 , a significance level of 0.05 , a 95% CI with its two sides of 0.112 and 0.46, the required sample size will be of 26 subjects that will undergo to bowel resection that must be associated with other 26 subjects with no bowel resection and other 26 will undergo delayed bowel resection, for a total of 78 patients. According to this sample size the score will have a sensitivity of 0.28, a specificity of 0.73, a positive predictive value of 0.22, a negative predictive value of 0.73 and a precision value of 0.39.

The optimal cut-off point with the highest sum of sensitivity and specificity will be chosen for each variable, also the overall predictive value of the Score will be assessed. Finally, a score will be developed by assigning coefficient points to each variable.

ELIGIBILITY:
Inclusion Criteria:

* All centers that routinely perform emergency laparoscopic surgery for SBO and have imaging systems with technology for the detection of near-infrared/indocyanine green fluorescence
* All patients more than 18 years old undergoing emergency laparoscopic surgery for SBO with intraoperative doubts about bowel viability after the resolution of the occlusive mechanism

Exclusion Criteria:

* Open surgical procedure for SBO

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients more undergoing emergency laparoscopic surgery for SBO with intraoperative doubts about bowel viability after the resolution of the occlusive mechanism
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Development of a resectability laparoscopic score based on data of a multicentric data registry | Event occurred at the time of surgery or after the first surgical interventional without bowel resection
  Based on these items a resectability laparoscopic score is developed:
  * Length of compromised bowel expressed in centimeters
  * Quality of peritoneal fluid
  * Time to presence of peristalsis after resolution of the obstruction expressed in minutes
  * Time of return to healty bowel coloration after resolution of the obstruction expressed in minutes
  * ICG-fluorescence angiographic patterns
  * Bowel resection rate expressed as event/non event
  * Reintervention rate expressed as event/non event
  * Date of reintervention expressed in days
  * Delayed bowel resection rate expressed as event/non event

SECONDARY OUTCOMES:
Development of a multicentric data registry of patients underwent laparoscopic approach to small bowel obstruction and ICG fluorescent angiography | 12 months eventually extended by further 6 months
  A Data Registry is constructed from multicentric data

CONTACTS AND LOCATIONS:
Overall Officials: DIEGO COLETTA, MD, Principal Investigator — San Salvatore Hospital, AST Pesaro-Urbino
Locations (1):
- Department of General Surgery, San Salvatore Hospital , AST Pesaro-Urbino, Pesaro, Pesaro-Urbino, Italy

IPD SHARING:
Plan to Share IPD: No